CLINICAL TRIAL: NCT05643417
Title: A Single Center, Multi Cohort, Phase I Basket Trial of the Safety and Efficacy of Camrelizumab in Combination With Bevacizumab and HAIC for Metastatic Liver Cancer After Standard Treatment Failure
Brief Title: Camrelizumab Combined With Bevacizumab and HAIC in Patients With Metastatic Liver Cancer Who Failed Standard Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-OBU-SH-CA-II-019
Record Dates: First submitted 2022-11-20; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Metastatic Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Liver metastasis of gastric cancer (Experimental): HAIC: refer to genetic test results，D1； Bevacizumab：7.5mg/Kg, D2, Q3W；Camrelizumab：200mg, D2, Q3W；
  Interventions: Drug: HAIC、Bevacizumab、Camrelizumab
- Liver metastasis of breast cancer (Experimental): HAIC: refer to genetic test results，D1；Bevacizumab：7.5mg/Kg, D2, Q3W；Camrelizumab：200mg, D2, Q3W；
  Interventions: Drug: HAIC、Bevacizumab、Camrelizumab
- Liver metastasis of lung cancer (Experimental): HAIC: refer to genetic test results，D1；Bevacizumab：7.5mg/Kg, D2, Q3W；Camrelizumab：200mg, D2, Q3W；
  Interventions: Drug: HAIC、Bevacizumab、Camrelizumab
- Liver metastasis of nasopharyngeal carcinoma (Experimental): HAIC: refer to genetic test results，D1；Bevacizumab：7.5mg/Kg, D2, Q3W；Camrelizumab：200mg, D2, Q3W；
  Interventions: Drug: HAIC、Bevacizumab、Camrelizumab
- Liver metastasis of thyroid cancer (Experimental): HAIC: refer to genetic test results，D1；Bevacizumab：7.5mg/Kg, D2, Q3W；Camrelizumab：200mg, D2, Q3W；
  Interventions: Drug: HAIC、Bevacizumab、Camrelizumab
- Liver metastasis of melanoma (Experimental): HAIC: refer to genetic test results，D1；Bevacizumab：7.5mg/Kg, D2, Q3W；Camrelizumab：200mg, D2, Q3W；
  Interventions: Drug: HAIC、Bevacizumab、Camrelizumab
- Liver metastasis of stromal tumor (Experimental): HAIC: refer to genetic test results，D1；Bevacizumab：7.5mg/Kg, D2, Q3W；Camrelizumab：200mg, D2, Q3W；
  Interventions: Drug: HAIC、Bevacizumab、Camrelizumab
- Liver metastasis of sarcoma (Experimental): HAIC: refer to genetic test results，D1；Bevacizumab：7.5mg/Kg, D2, Q3W；Camrelizumab：200mg, D2, Q3W；
  Interventions: Drug: HAIC、Bevacizumab、Camrelizumab
- Liver metastasis of other solid tumor (Experimental): HAIC: refer to genetic test results，D1；Bevacizumab：7.5mg/Kg, D2, Q3W；Camrelizumab：200mg, D2, Q3W；
  Interventions: Drug: HAIC、Bevacizumab、Camrelizumab

INTERVENTIONS:
Drug: HAIC、Bevacizumab、Camrelizumab — HAIC: refer to genetic test results，D1 Bevacizumab：7.5mg/Kg, D2, Q3W Camrelizumab：200mg, D2, Q3W
  Other Names: Camrelizumab brand name: ai rui ka; Bevacizumab brand name: ai rui tuo

SUMMARY:
This is a single center, multi-cohort, phase I basket trial to evaluate the safety and efficacy of camrelizumab in combination with bevacizumab and HAIC for metastatic liver cancer after standard treatment failure

DETAILED DESCRIPTION:
For patients with advanced primary liver cancer, immunotherapy combined anti-angiogenic therapy has gradually become the first-line standard treatment. However, for metastatic liver cancer, especially after first-line treatment failure, the current treatment options are mostly systemic chemotherapy, and there is still a lack of effective treatment methods. Compared with systemic chemotherapy, HAIC has a higher objective response rate and survival rate, and the incidence of adverse reactions is lower. At the same time, PD-1 combined with chemotherapy has become the first-line standard treatment for many cancers; referring to the expert consensus on liver metastasis of solid tumors and ongoing clinical research, the "PD-1 + anti-angiogenesis + HAIC" regimen can be used as a new research direction for posterior treatment for metastatic liver cancer.

In view of the failure of first-line chemotherapy, how to find effective chemotherapy drugs has become a top priority. HAIC guided by genetic testing may be able to screen out effective chemotherapy drugs

This study is an open-label, single-center, multi-cohort, phase I basket trial designed to explore safety and efficacy of "camrelizumab + bevacizumab + HAIC guided by genetic testing" for metastatic liver cancer after standard treatment failure

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been signed
2. Age ≥ 18 years old
3. Liver metastases of solid tumors confirmed by histology or cytology (including but not limited to gastric cancer, breast cancer, lung cancer, nasopharyngeal cancer, thyroid cancer, melanoma, stromal tumor, sarcoma, etc.), including liver metastases at the time of diagnosis or liver metastases occurred after radical resection, and the primary tumor has been resected
4. The investigator assessed that the liver metastasis could not be removed surgically
5. Progression or intolerance after receiving standard systemic therapy (patients who have received first-line immunotherapy can still be enrolled)
6. Child-Pugh score ≤ 7
7. At least one measurable lesion (according to RECIST 1.1)
8. Expected overall survival ≥ 3 months
9. ECOG PS score: 0~1
10. Has sufficient organ function within 14 days before the first administration, (1) Blood routine: WBC≥3.0×109/L; ANC≥1.5×109/L; PLT≥50×109/L; HGB≥90 g/L (2) Liver function: AST≤5.0×ULN; ALT≤5.0×ULN; TBIL≤2.0×ULN (3) Renal function: Cr≤1.5×ULN or CrCl ≥60 mL/min (4) Coagulation function: INR≤1.5; APTT≤1.5×ULN (5) HBV-DNA≤2×103 IU/ml (subjects with HBV-DNA>2×103 IU/ml can be enrolled and should receive antiviral treatment at the same time)
11. Women of childbearing age must take contraceptive measures within 3 months from the first dose to the last use of the study drug

Exclusion Criteria:

1. Patients had other malignant tumors in the past or at the same time (excluding non melanoma skin cancer, cervical carcinoma in situ, papillary thyroid cancer after treatment)
2. Patients had a history of organ transplantation or hepatic encephalopathy
3. Suffering from immunodeficiency disease within 7 days before the first administration, or receiving systemic hormone treatment (≥ 10mg/day prednisone or equivalent dose of other hormones), or other forms of immunosuppressive treatment
4. Patients who are seriously allergic to iodized contrast agents, antibody drugs, calcium folinate, 5-FU, platinum drugs , (≥ grade 3)
5. Participated in other clinical trials or received other test drugs within 4 weeks before the first administration
6. Pregnant or lactating women or women of childbearing age are positive in the baseline pregnancy test
7. Other factors that may affect the subject's safety or test compliance as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and degree of Adverse Events and Serious Adverse Events | 24 months
  Incidence, severity, and relationship to study drugs of all adverse events (AEs), treatment-related adverse events (TRAEs), and serious adverse events (SAEs).
ORR | 24 months
  objective response rate(ORR)，defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.

SECONDARY OUTCOMES:
DCR | 24 months
  disease control rate(DCR), defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
PFS | 24 months
  progression-free survival(PFS), defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
OS | 24 months
  overall survival(OS), defined as the time from enrollment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Wang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China